CLINICAL TRIAL: NCT04259502
Title: Comparison of Rhomboid Intercostal Block and Erector Spina Plan Block for Peri-operative Analgesia in Mastectomy
Brief Title: Rhomboid Intercostal Block vs Erector Spina Plan Block for Peri-operative Analgesia in Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Onur Balaban, MD, Asistan Professor, MD., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/06RIBVSESP
Record Dates: First submitted 2020-01-13; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Analgesia; Perioperative Analgesia; Postoperative Analgesia
Keywords: Postoperative Analgesia; Peroperative Analgesia; Ultrasound; Rhomboid intercostal block; Erector spinae plane block; Mastectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The patients included in the study will be assigned to one group of two in which two different regional block technique will be performed alone.
Who Masked: Participant, Care Provider
Masking Description: The two interventions will be performed at the same thoracic region using the same technique as so; there participant will be blinded to the study. The investigator who performs the intervention will be unblinded. The investigator who will follow up the patients and collect the postoperative pain data will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIB Group (Experimental): A single injection Rhomboid intercostal block will be performed under ultrasound guidance
  Interventions: Procedure: Rhomboid intercostal block
- ESP Group (Active Comparator): A single injection Erector spinae plane block will be performed under ultrasound guidance
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Rhomboid intercostal block — The block is regional anesthesia injection techniques performed under ultrasound guidance.
  Arms: RIB Group
Procedure: Erector spinae plane block — The block is regional anesthesia injection techniques performed under ultrasound guidance.
  Arms: ESP Group

SUMMARY:
Effectiveness of erector spinae plane block for analgesia in breast surgery was documented in previous studies. Rhomboid intercostal block may be beneficial for analgesia in breast surgery. The aim of this study is to compare the peri-operative analgesic effect of rhomboid intercostal block with erector spinae plane block in mastectomy operation. This trial was designed as prospective randomized single-blind study. The included patients will be assigned into two groups: RIB-Group where the patients will receive ultrasound-guided rhomboid intercostal block and ESP-Group where the patients will receive ultrasound-guided erector spinae plane block prior to the operation. Primary outcome will be peri-operative pain scores and secondary outcomes will be peri-operative opioid consumption and peri-operative hemodynamic effect of these blocks.

DETAILED DESCRIPTION:
Postoperative analgesia in breast surgery is important in reducing morbidity and mortality. Intravenous or oral analgesics may be used for this purpose. Ultrasound-guided fascia plane blocks are used to provide effective analgesia in mastectomy operations. Effectiveness of erector spinae plane block for analgesia in breast surgery was documented in previous studies.

Rhomboid intercostal block may be beneficial for analgesia in breast surgery. Both blocks have the advantage of unilateral application in unilateral mastectomy operations. When administered pre-operatively, it also provides per-operative analgesia and may reduce per-operative opioid consumption. These blocks are applied under ultrasound-guidance with single injection. Since the site of injection is relatively superficial (between the back muscles and ribs) and applied under ultrasound-guidance, mechanical complications is expected to occur less. These low-cost blocks also may reduce the usage of high-cost and high-risk opioids after surgery. These blocks unilaterally anesthetize the nerves innervating the thoracic region and the axilla, thus providing effective per-operative and post-operative analgesia in mastectomy operations.

The aim of our study is to compare the rhomboid intercostal block with erector spina plane block in mastectomy in terms of intraoperative and postoperative analgesia in mastectomy operation. Our hypothesis is rhomboid intercostal block may reduce peri-operative pain as effective as or more effectively than erector spina plane block. Secondary hypothesis is rhomboid intercostal block may reduce peri-operative opioid consumption as effective as or more effectively than erector spina plane block. Thus, the study is defined as block technique comparison.

Eighty patients aged between 29-79 years who are planned mastectomy under general anesthesia will be included in the study. Patients with severe cardiac and respiratory disease, severe coagulation disorder, body mass index greater than 35, refusal of regional block and patients having local infection in block application area, contraindication of the standardized drugs in the study and patients with insufficient postoperative analgesia requiring more potent opioids will be excluded from the study.

The patients who meet the study criteria will be assigned into two groups by using computerized randomization. Patients who do not give consent will also be excluded from the study. All patients will be sedated with midazolam and fentanyl prior to block application. First group (RIB-Group) of patients will receive ultrasound-guided rhomboid intercostal block prior to the operation under sedation. Patients in the second group (ESP-Group) will receive ultrasound-guided erector spina plane block under sedation. Since both procedures will be performed from the same site, the study was considered as a single blind.

All patients will be intubated after induction of general anesthesia with Propofol 2 mg / kg, Rocuronium 0.6 mg / kg and Fentanyl 1.5 µg / kg. Mixture of Desflurane 6% concentration in 50% air and 50% oxygen will be used for the maintenance of general anesthesia. Patients in both groups will receive 1 µg / kg of fentanyl when pain occurs during surgery. Pre-operative and post-operative blood pressure, heart rate, oxygen saturation, end-tidal carbon dioxide values of patients in both groups will be measured and recorded at determined time intervals.

Patients will be followed for 48 hours after the operation. In the postoperative period, acetaminophen 1 g three times a day will be administered routinely in context of multimodal analgesia. Intravenous tramadol 1 mg/kg will also be administered depending on patient need up to 4 times a day. Total amount of perioperative opioids will be recorded. Per-operative and post-operative opioid consumption will be calculated separately. Pain assessment will be evaluated by using a verbal analog scale (asking patients to give a pain score between 0 and 10. Score of 0 means worse pain ever and score of 10 means no pain). Complications related to the block procedure will be also recorded. If there is pain that requires more potent opioids such as morphine, the block will be considered as unsuccessful.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned mastectomy under general anesthesia

Exclusion Criteria:

* Patients with severe cardiac and respiratory disease
* Severe coagulation disorder
* Body mass index greater than 35 kg/m2
* Refusal of regional block
* Patients having local infection in block application area
* Contraindication of the standardized drugs in the study
* Insufficient postoperative analgesia requiring more potent opioids

Ages: 29 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Pain score | Throughout post-operative course, up to 48 hours
  Subjective pain score reported by the patient, assessed by a blinded investigator to the study; which is defined as the score in a scale between minimum value of zero and maximum value of 10 (higher scores mean a better outcome).
Peroperative Analgesia | At the end of the operation
  Fentanyl consumption

SECONDARY OUTCOMES:
Opioid consumption | 48th postoperative hour
  Total tramadol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Onur Balaban, MD., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elsharkawy H, Saifullah T, Kolli S, Drake R. Rhomboid intercostal block. Anaesthesia. 2016 Jul;71(7):856-7. doi: 10.1111/anae.13498. No abstract available. PMID 27291611
- [Background] Balaban O, Aydin T. A modified approach of rhomboid intercostal block for postoperative analgesia in modified radical mastectomy: Ultrasound guided bi-level high thoracic injection. J Clin Anesth. 2019 Nov;57:29-30. doi: 10.1016/j.jclinane.2019.03.002. Epub 2019 Mar 6. No abstract available. PMID 30851500
- [Background] Yayik AM, Ahiskalioglu A, Ates I, Ahiskalioglu EO, Cinal H. Ultrasound guided bilateral rhomboid intercostal block for breast reduction surgery. J Clin Anesth. 2019 Nov;57:38-39. doi: 10.1016/j.jclinane.2019.03.001. Epub 2019 Mar 6. No abstract available. PMID 30851503
- [Background] Tulgar S, Selvi O, Thomas DT, Manukyan M, Ozer Z. Rhomboid intercostal block in a modified radical mastectomy and axillary curettage patient; A new indication for novel interfascial block. J Clin Anesth. 2019 May;54:158-159. doi: 10.1016/j.jclinane.2018.12.006. Epub 2018 Dec 13. No abstract available. PMID 30553225
- [Background] Singh S, Kumar G, Akhileshwar. Ultrasound-guided erector spinae plane block for postoperative analgesia in modified radical mastectomy: A randomised control study. Indian J Anaesth. 2019 Mar;63(3):200-204. doi: 10.4103/ija.IJA_758_18. PMID 30988534
- [Background] Selvi O, Tulgar S. Use of the Ultrasound-Guided Erector Spinae Plane Block in Segmental Mastectomy. Turk J Anaesthesiol Reanim. 2019 Apr;47(2):158-160. doi: 10.5152/TJAR.2019.50024. Epub 2019 Jan 29. PMID 31080959
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Kimachi PP, Martins EG, Peng P, Forero M. The Erector Spinae Plane Block Provides Complete Surgical Anesthesia in Breast Surgery: A Case Report. A A Pract. 2018 Oct 1;11(7):186-188. doi: 10.1213/XAA.0000000000000777. PMID 29688930
- [Background] Aksu C, Kus A, Yorukoglu HU, Tor Kilic C, Gurkan Y. Analgesic effect of the bi-level injection erector spinae plane block after breast surgery: A randomized controlled trial. Agri. 2019 Jul;31(3):132-137. doi: 10.14744/agri.2019.61687. PMID 31736025
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Turan M, Gumus Demirbilek S. Comparison of the effects of modified pectoral nerve block and erector spinae plane block on postoperative opioid consumption and pain scores of patients after radical mastectomy surgery: A prospective, randomized, controlled trial. J Clin Anesth. 2019 May;54:61-65. doi: 10.1016/j.jclinane.2018.10.040. Epub 2018 Nov 3. PMID 30396100
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH. Erector spinae plane block and thoracic paravertebral block for breast surgery compared to IV-morphine: A randomized controlled trial. J Clin Anesth. 2020 Feb;59:84-88. doi: 10.1016/j.jclinane.2019.06.036. Epub 2019 Jul 4. PMID 31280100